CLINICAL TRIAL: NCT03829748
Title: Intermittent Versus Continuous Suction Technique in the Diagnosis of Pancreatic Solid Lesions. A Pilot Study.
Brief Title: Intermittent Suction Technique in the Diagnosis of Pancreatic Solid Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: RHerranz3638
Record Dates: First submitted 2019-01-22; First posted 2019-02-04 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Pancreatic Cancer; Pancreatic Neoplasms
Keywords: Pancreatic adenocarcinoma; Endoscopic ultrasound; Fine-needle aspiration
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent aspiration (Experimental): Empty syringe of 10cc and intermittent aspiration during puncture
  Interventions: Procedure: Intermittent aspiration
- Continous/standard aspiration (No Intervention): Empty syringe of 10cc and continous aspiration during puncture

INTERVENTIONS:
Procedure: Intermittent aspiration — Endoscopic ultrasound is done for the localization of the lesion and to localize the site of puncture.Prior to the puncture of the lesion the stylet is removed and a vacuum syringe is prepared with 10 cc of vacuum allowing the generation of continous pressure inside and connected to the end of the needle. Once the lesion is punctured 15 movements in and out of the lesions will be made while the syringe is opened and closed on and off for a total of 3 times each pass. A total of 4 passes will be done in each lesion.
  Arms: Intermittent aspiration

SUMMARY:
The aim of this study is to compare the diagnostic yield of intermittent versus continuous suction in the diagnosis of pancreatic solid lesions.

DETAILED DESCRIPTION:
Solid lesions of the pancreas can be neoplastic or non neoplastic and it is important to accurately differentiate between them because of the poor prognosis related to pancreatic neoplasm. There are many types of solid pancreatic lesions: pancreatic adenocarcinoma, neuroendocrine tumor, lymphoma, solid pseudopapillary neoplasm and pancreatic metastasis.

There are several diagnostic methods for the study of pancreatic solid lesions. The different imaging test allow detection and characterization of those lesions, but most times an anatomopathological diagnosis is needed before stablishing the most appropriate treatment.

Endoscopic Ultrasound guided fine needle aspiration (EUS-FNA) is the diagnostic method of choice for the diagnosis of these lesions as it detects small lesions that sometimes cannot be found in radiological imaging test, evaluates vascular invasion and the presence of liver metastasis, and allows pancreatic puncture for a cytological diagnosis. EUS-FNA is the safest technique for pancreatic puncture and the least related to needle track seeding.

In order to gather as much material as possible different techniques have been proposed:

* Fanning technique and multiple pass technique: to guide the needle into different regions of the target lesions with or without removing the needle out of the lesion depending on wether the lesion is hard or soft.
* Use of stylet: there are no data clearly demonstrating that the use of suction increases the yield of EUS-FNA. Some authors do slow withdrawal of the stylet.
* Size of the needle: 19 gauge, 22 gauge, 25 gauge, depending on the localization, size and vascularization. There is increasing evidence that smaller needles offer at least similar results in diagnostic yield compared to larger needles and are also easier to manipulate.
* Use of suction: there is conflicting evidence in this point. Several studies have evaluated the use of high volume aspiration vs low volume aspiration, continous aspiration vs no aspiration and suction with empty syringe vs water-filled syringe but none is clearly better than other.

The investigators aim is to evaluate if the use of intermittent suction improves the diagnostic yield of pancreatic lesions compared to standard (continuous) suction. Up to our knowledge this method has not been yet evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic solid lesion
* Patients over 18 years old
* Suitable for endoscopy

Exclusion Criteria:

* Contraindication for endoscopy
* Active anticoagulant therapy
* Thrombocytopenia or coagulopathy in the absence of its correction prior to the procedure
* Absence of informed consent
* Pregnancy
* Not accessible lesion for endoscopic ultrasound puncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Increase in diagnostic yield of pancreatic solid lesions | Baseline
  Percentage of increase in positive smears between intermittent and continous suction

SECONDARY OUTCOMES:
Sample cellularity | Baseline
  Number of malignant clusters of cells on each endoscopic pass
Blood contamination | Baseline
  Percentage of blood contamination of the slides
Number of passes to reach diagnosis | Baseline
  Number of passes needed to achieve a positive cytological diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Herranz Pérez, MD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (1):
- Hospital Universitario de la Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT03829748/Prot_SAP_001.pdf